CLINICAL TRIAL: NCT01610232
Title: Effects of Infrared-LED Illumination Applied During Treadmill Training in Postmenopausal Women
Brief Title: Infrared-LED During Physical Training for Rehabilitation, Physical Performance and Body Aesthetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Fernanda Rossi Paolillo, Ph.D, University of Sao Paulo
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 98142708
Record Dates: First submitted 2012-05-30; First posted 2012-06-01 (Estimated); Last update posted 2012-06-01 (Estimated); Status verified 2012-05

CONDITIONS: Healthy
Keywords: Infrared LED; Treadmill Training; Strength Muscle; Fatigue Muscle; Aerobic Capacity; Cellulite; Osteoporosis
MeSH Terms: conditions — Cellulite; Osteoporosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- LED Group (Experimental): Phototherapy associated with treadmill training
  Interventions: Device: Photon stimulation by light-emitting diodes (LEDs)
- Exercise Group (Active Comparator): Treadmill training
  Interventions: Other: Treadmill training
- Sedentary Group (No Intervention): Neither physical training nor phototherapy

INTERVENTIONS:
Device: Photon stimulation by light-emitting diodes (LEDs) — Treadmill training with the application of the phototherapy was performed twice a week for 6 months, each session lasting 45 min at intensities between 85% and 90% maximal heart rate. The average power and power density on the skin were 100 mW and 39 mW/cm2, respectively. The treatment time was 45 min bilaterally in both thighs. These parameters led to an approximate fluence of 108 J/cm2.
  Arms: LED Group
Other: Treadmill training — Treadmill training without the application of the phototherapy was performed twice a week for 6 months, each session lasting 45 min at intensities between 85% and 90% maximal heart rate
  Arms: Exercise Group

SUMMARY:
The investigators hypothesis is that the infrared-LED illumination during treadmill training can enhance physical performance in postmenopausal women. The basis for such a hypothesis is based on the fact that the light therapy during the intense metabolic stage caused by exercise may be more efficient.

DETAILED DESCRIPTION:
Phototherapy improves cellular activation via absorption of photons by chromophores present in the protein components of the mitochondrial respiratory chain - mainly NADH dehydrogenases and cytochrome C oxidase, which leads to increased electron transport, production of ATP, and tissue regeneration (skin, muscle, bone, and nerves). Moreover, phototherapy stimulates the anti-inflammatory effect with analgesia and vasodilatation. Regarding body aesthetics, phototherapy increases microcirculation, lymphatic drainage, as well as collagen synthesis for the treatment of cellulite. The objective of this study was to develop and evaluate the effects of a new clinical procedure: infrared radiation originated from LEDs associated with treadmill training in postmenopausal women. LED arrays were developed for an irradiation of a large area, such as hip and quadriceps muscles, main actuators during stance and swing phases. These body parts are furthermore areas where there is incidence of osteoporosis, mainly at the femur, localized fat deposits, and cellulite. Infrared radiation (850 nm) was selected because this spectral range shows better skin penetration compared to red interval.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women
* Caucasian
* 50 and 60 years of age
* Healthy

Exclusion Criteria:

* Neurological disease
* Inflammatory disease
* Pulmonary disease
* Oncological disease
* Cardiac disease
* Endocrinopathy
* Musculotendinous or articular injuries
* Hormone replacement therapy or osteoporosis drugs
* Cigarette smoking

Ages: 50 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2009-12; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Effects of Infrared-LED Illumination Associated with Treadmill Training | 12 months
  Quantitative and qualitative evaluations

SECONDARY OUTCOMES:
Maximal exercise testing | Baseline and 6 months
  Progressive aerobic exercise testing on treadmill (Modified Bruce Protocol)
Isokinetic concentric exercise testing | Baseline, 6 months and 12 months
  Peak torque, power, work, and fatigue of the dominant quadriceps were measured using the isokinetic dynamometer
Biochemical tests | Baseline and 6 months
  Thyroid stimulating hormone (TSH), urea, creatinine, triglycerides, total cholesterol, high-density lipoprotein (HDL) cholesterol, low-density lipoprotein (LDL) cholesterol, very low-density lipoprotein (VLDL) cholesterol, insulin and glucose
Quality of life | Baseline and 6 months
  Menopause Rating Scale (MRS) and Women´s Health Questionnaire (WHQ)
Dietary habits | Baseline and 6 months
  3-day dietary record
Exercise tolerance and heart rate variability | Baseline and 6 months
  Submaximal constant-speed testing and heart rate variability via autonomic reflex testing
Bone mineral density | Baseline and 12 months
  Bone mineral density (femoral neck, wrist, and lumbar spine) via dual-energy x-ray absorptiometry (DXA)
Thermography | Baseline
  Cutaneous temperature measurements

CONTACTS AND LOCATIONS:
Overall Officials: Vanderlei S Bagnato, Ph.D, Study Director — Physics Institute of São Carlos (IFSC), University of São Paulo (USP); Cristina Kurachi, Ph.D, Study Director — Physics Institute of São Carlos (IFSC), University of São Paulo (USP); Fernanda R Paolillo, Ph.D, Principal Investigator — Physics Institute of São Carlos (IFSC), University of São Paulo (USP)
Locations (1):
- Optics Group from Physics Institute of São Carlos (IFSC), University of São Paulo (USP), São Carlos, São Paulo, Brazil

REFERENCES:
- [Background] Ferraresi C, de Brito Oliveira T, de Oliveira Zafalon L, de Menezes Reiff RB, Baldissera V, de Andrade Perez SE, Matheucci Junior E, Parizotto NA. Effects of low level laser therapy (808 nm) on physical strength training in humans. Lasers Med Sci. 2011 May;26(3):349-58. doi: 10.1007/s10103-010-0855-0. Epub 2010 Nov 18. PMID 21086010
- [Background] Vieira WH, Ferraresi C, Perez SE, Baldissera V, Parizotto NA. Effects of low-level laser therapy (808 nm) on isokinetic muscle performance of young women submitted to endurance training: a randomized controlled clinical trial. Lasers Med Sci. 2012 Mar;27(2):497-504. doi: 10.1007/s10103-011-0984-0. Epub 2011 Aug 26. PMID 21870127
- [Background] De Marchi T, Leal Junior EC, Bortoli C, Tomazoni SS, Lopes-Martins RA, Salvador M. Low-level laser therapy (LLLT) in human progressive-intensity running: effects on exercise performance, skeletal muscle status, and oxidative stress. Lasers Med Sci. 2012 Jan;27(1):231-6. doi: 10.1007/s10103-011-0955-5. Epub 2011 Jul 8. PMID 21739259
- [Background] Baroni BM, Leal Junior EC, Geremia JM, Diefenthaeler F, Vaz MA. Effect of light-emitting diodes therapy (LEDT) on knee extensor muscle fatigue. Photomed Laser Surg. 2010 Oct;28(5):653-8. doi: 10.1089/pho.2009.2688. Epub 2010 Jul 13. PMID 20626264
- [Background] Leal Junior EC, Lopes-Martins RA, Baroni BM, De Marchi T, Rossi RP, Grosselli D, Generosi RA, de Godoi V, Basso M, Mancalossi JL, Bjordal JM. Comparison between single-diode low-level laser therapy (LLLT) and LED multi-diode (cluster) therapy (LEDT) applications before high-intensity exercise. Photomed Laser Surg. 2009 Aug;27(4):617-23. doi: 10.1089/pho.2008.2350. PMID 19302015
- [Background] Karu TI, Pyatibrat LV, Afanasyeva NI. Cellular effects of low power laser therapy can be mediated by nitric oxide. Lasers Surg Med. 2005 Apr;36(4):307-14. doi: 10.1002/lsm.20148. PMID 15739174
- [Background] Corazza AV, Jorge J, Kurachi C, Bagnato VS. Photobiomodulation on the angiogenesis of skin wounds in rats using different light sources. Photomed Laser Surg. 2007 Apr;25(2):102-6. doi: 10.1089/pho.2006.2011. PMID 17508845
- [Background] Whelan HT, Smits RL Jr, Buchman EV, Whelan NT, Turner SG, Margolis DA, Cevenini V, Stinson H, Ignatius R, Martin T, Cwiklinski J, Philippi AF, Graf WR, Hodgson B, Gould L, Kane M, Chen G, Caviness J. Effect of NASA light-emitting diode irradiation on wound healing. J Clin Laser Med Surg. 2001 Dec;19(6):305-14. doi: 10.1089/104454701753342758. PMID 11776448
- [Background] Vladimirov YA, Osipov AN, Klebanov GI. Photobiological principles of therapeutic applications of laser radiation. Biochemistry (Mosc). 2004 Jan;69(1):81-90. doi: 10.1023/b:biry.0000016356.93968.7e. PMID 14972023
- [Result] Paolillo FR, Milan JC, Aniceto IV, Barreto SG, Rebelatto JR, Borghi-Silva A, Parizotto NA, Kurachi C, Bagnato VS. Effects of infrared-LED illumination applied during high-intensity treadmill training in postmenopausal women. Photomed Laser Surg. 2011 Sep;29(9):639-45. doi: 10.1089/pho.2010.2961. Epub 2011 Jul 12. PMID 21749263
- [Result] Paolillo FR, Borghi-Silva A, Parizotto NA, Kurachi C, Bagnato VS. New treatment of cellulite with infrared-LED illumination applied during high-intensity treadmill training. J Cosmet Laser Ther. 2011 Aug;13(4):166-71. doi: 10.3109/14764172.2011.594065. PMID 21740089
- [Result] Paolillo FR, Corazza AV, Borghi-Silva A, Parizotto NA, Kurachi C, Bagnato VS. Infrared LED irradiation applied during high-intensity treadmill training improves maximal exercise tolerance in postmenopausal women: a 6-month longitudinal study. Lasers Med Sci. 2013 Feb;28(2):415-22. doi: 10.1007/s10103-012-1062-y. Epub 2012 Mar 2. PMID 22382875
- [Result] Paolillo FR, Milan JC, Bueno Pde G, Paolillo AR, Borghi-Silva A, Parizotto NA, Arena R, Kurachi C, Bagnato VS. Effects of excess body mass on strength and fatigability of quadriceps in postmenopausal women. Menopause. 2012 May;19(5):556-61. doi: 10.1097/gme.0b013e3182364e80. PMID 22089183
- See also: Research: Biophotonics (phototherapy) — http://cepof.ifsc.usp.br/